CLINICAL TRIAL: NCT06759246
Title: Short Implant Placement for Single-Tooth Rehabilitation in the Atrophic Posterior Maxilla
Brief Title: Short Implants in Atrophic Posterior Maxilla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Giuseppe D'Albis, Dr. D'Albis Giuseppe, University of Bari Aldo Moro
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Implants01
Record Dates: First submitted 2024-11-15; First posted 2025-01-06 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Edentulism; Bone Atrophy, Alveolar; Sinus Pneumatization
Keywords: short implants; bone atrophy; sinus pneumatization; minimal invasive
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atrophic maxillae (Other): A group of patients with atrophic maxillae requiring rehabilitation for single-tooth edentulism.
  Interventions: Procedure: implant placement

INTERVENTIONS:
Procedure: implant placement — Placement of short implants for the rehabilitation of single-tooth edentulism in atrophic maxillae near the maxillary sinus.

SUMMARY:
This study aims to evaluate the clinical and radiological outcomes of short implants in the rehabilitation of single-tooth edentulism in the posterior maxilla. By assessing these outcomes, the research seeks to determine the effectiveness and long-term viability of short implants as a minimally invasive solution, particularly in cases where bone height is limited.

DETAILED DESCRIPTION:
The present municentric retrospective study was conducted following the STROBE statement recommendations for observational studies and in compliance to the principles of the Declaration of Helsinki on clinical research involving human subjects.The study aims to evaluate short implants placed over the past 15 years by three experienced clinicians, assessing their survival and clinical success. Specifically, the study collects clinical data such as probing depth, the presence or absence of peri-implantitis, and radiological findings.

ELIGIBILITY:
Inclusion Criteria:

* Good health status according to the classification system of the American Society of Anesthesiology (ASA), and patients were required to be 18 years of age or older.
* No general medical condition that would contraindicate implant therapy.
* No active periodontal disease, defined as a periodontal probing depth of less than 4 mm, or previously treated periodontitis.
* Good oral hygiene, with a full-mouth plaque index of less than 25%.
* Adequate control of inflammation, with a full-mouth bleeding on probing (BOP) of less than 25%.

Exclusion Criteria:

* Smoking more than 15 cigarettes per day
* Presence of untreated periodontal disease
* Pregnancy or breastfeeding at the time of enrollment
* Active infections
* Less than 2 mm of keratinized mucosal tissue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Clinical outcome | 2 years
  Survival rate: A statistical analysis will be conducted to evaluate the implant survival rate at three specific time points: T1 (3 months), T2 (6 months), and T3 (2 years).

SECONDARY OUTCOMES:
Rx outcome | 2 years
  Radiographic measurements will be obtained using standardized imaging techniques. The measurements will be performed digitally using dedicated three-dimensional radiological imaging software, ensuring high precision. Distances will be measured in millimeters to evaluate implant positioning, bone levels, and defect morphology with accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Saverio Capodiferro, Study Director — University of Bari Aldo Moro; Professor Massimo Corsalini, Study Director — University of Bari Aldo Moro; Dr. D'Albis Giuseppe, Principal Investigator — University of Bari Aldo Moro
Locations (1):
- University of Bari Aldo Moro, Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Corsalini M, D'Agostino S, Favia G, Dolci M, Tempesta A, Di Venere D, Limongelli L, Capodiferro S. A Minimally Invasive Technique for Short Spiral Implant Insertion with Contextual Crestal Sinus Lifting in the Atrophic Maxilla: A Preliminary Report. Healthcare (Basel). 2020 Dec 24;9(1):11. doi: 10.3390/healthcare9010011. PMID 33374157